CLINICAL TRIAL: NCT01019408
Title: Clinical Trial of Extended-dose Chloroquine Versus Standard Chloroquine Treatment for Resistant Falciparum Malaria Among Afghan Refugees in NWFP Pakistan
Brief Title: Extended-dose Chloroquine (ECQ) for Resistant Falciparum Malaria Among Afghan Refugees in Pakistan
Acronym: ECQNWFP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: European Union (Other); United Nations High Commissioner for Refugees (Other); World Health Organization (Other)
Responsible Party: Mark Rowland, LSHTM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-HNI01
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Malaria, Falciparum
Keywords: Clinical Trial; Chloroquine; Refugees; Afghanistan; Pakistan
MeSH Terms: conditions — Malaria, Falciparum | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CQ25 (Active Comparator): Falciparum positive patients receiving standard 3-day treatment course of CQ 25mg/kg.
  Interventions: Drug: Chloroquine
- CQ40 (Active Comparator): Falciparum positive patients receiving a 5-day treatment course of CQ 40 mg/kg.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — Comparison of two different dosages of chloroquine for treatment of falciparum malaria in Afghan refugee camps in Northwest Frontier Province, Pakistan
  Other Names: CQ

SUMMARY:
The purpose of this study was to provide stronger evidence for extended-dose chloroquine treatment of falciparum-positive Afghan refugees in Northwest Frontier Province (NWFP), Pakistan or justification for discontinuation of the policy.

DETAILED DESCRIPTION:
To determine whether extended-dose chloroquine provided better cure rates and fewer recrudescences than standard chloroquine treatment among Afghan refugees, 163 falciparum patients from three Afghan refugee camps were recruited into 3-day (CQ 25mg/kg) or 5-day (CQ 40mg/kg) treatment arms and followed for up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

* slide-confirmed infection with P. falciparum only
* initial parasite density of 1000-100,000 asexual parasites/μl
* absence of severe malnutrition
* ability to attend stipulated follow-up visits and easy access to facility
* informed consent provided by patient or parent/guardian
* absence of history of hypersensitivity reactions to CQ

Exclusion Criteria:

* infants under six months old
* pregnancy or lactation
* underlying chronic severe illness
* patients with other febrile illnesses
* parasitaemia outside the range of 1000-100,000 asexual parasites/µl
* severe malaria

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 1993-11; Primary Completion 1995-01 (Actual); Study Completion 1995-01 (Actual)

PRIMARY OUTCOMES:
therapeutic and parasitological cure with no recrudescence | 60 days

SECONDARY OUTCOMES:
parasite clearance time | 28 days
fever clearance time | 28 days
gametocytaemia | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rowland, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (3):
- Pakistan (3):
  - Adezai Basic Health Unit, Adezai, Khyber Pakhtunkhwa
  - Baghicha Basic Health Unit, Bāghīcha, Khyber Pakhtunkhwa
  - Kagan Basic Health Unit, Kagan, Khyber Pakhtunkhwa